CLINICAL TRIAL: NCT00859950
Title: Mechanisms of Endothelial Cell Dysfunction in Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ana C. Krieger, Dr. Ana Krieger, MD. MPH, Weill Medical College of Cornell University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0811010102; 1K23HL094358-01A2 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea; Hypoxemia
Keywords: Sleep Apnea; Vascular Occlusion; Nocturnal Polysomnography; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypoxia; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep Apnea (Active Comparator): Subjects found to have Obstructive Sleep Apnea (OSA) with Intermittent Hypoxemia (IH). This arm will undergo a pre-treatment blood draw, one month of Continuous Positive Airway Pressure (CPAP) to treat OSA, and a post-treatment blood draw.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- Normal Control (No Intervention): Subject found to have no evidence of Obstructive Sleep Apnea (OSA) after Nocturnal Polysomnography (NPSG). These subjects will only undergo a blood draw and will not have the Continuous Positive Airway Pressure (CPAP) treatment.

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — Continuous positive airway pressure (CPAP) is a method of respiratory ventilation which is accepted as the gold standard to treat Obstructive Sleep Apnea (OSA). Subjects found to have OSA after the Nocturnal Polysomnography (NPSG) will be trained in the use of CPAP and will be instructed to use CPAP every night for 30 nights. These subjects will then return for a post-treatment blood draw.
  Arms: Sleep Apnea

SUMMARY:
Sleep apnea is a common sleep disorder characterized by temporary stops in breathing during sleep and has been associated with the development of cardiovascular disease. This research will investigate one potential mechanism leading to the development of cardiovascular disorder, specifically, the blockage of blood vessels called "vascular occlusion", in subjects with sleep apnea. A group of healthy controls will be used for comparison. All subjects will undergo clinical evaluation followed by an overnight sleep study and a morning blood draw. Subjects with sleep apnea will be treated according to standard clinical management and followed under the research protocol for one month. At the end of one month, a repeat blood draw will be performed on the sleep apnea subjects for comparative analysis. If a control subject is found to have any abnormality during this research study, he or she will be referred for further clinical evaluation.

DETAILED DESCRIPTION:
The importance of this project is to investigate mechanisms of vascular disease in sleep apnea and determine pathways for intervention, aiming to prevent the development of cardiovascular disease in these individuals.

This proposed research aims to evaluate both NTPDase activity in lymphocytes and levels of circulating endothelial cells (CECs) in patients with intermittent hypoxemia (IH) due to obstructive sleep apnea (OSA) and healthy controls. This is an original approach to define mechanisms which underlie the high incidence of occlusive vascular events in patients with OSA. The evaluation of such pathophysiological mechanisms will lead to a better understanding of the pathways involved and the development of therapeutic strategies targeting the reduction or avoidance of endothelial injury with the ultimate goal of reducing morbidity and mortality associated with these pathologic events in sleep apnea. The standard of care will be used in this protocol, which involves the use of CPAP (continuous positive airway pressure) for treating sleep apnea.

ELIGIBILITY:
Study Group 1: Sleep Apnea

Inclusion Criteria:

* 21 years or older
* Presence of intermittent hypoxemia (IH) and obstructive sleep apnea (OSA)
* No diagnosis of hypertension, coronary artery disease, diabetes, stroke, or evidence of underlying vascular disease

Exclusion Criteria:

* Smoking
* Pregnancy
* Known cardiovascular disease, stroke, or diabetes
* Current or previous treatment for sleep apnea
* Central or Cheyne-Stokes sleep apnea
* Use of supplemental oxygen at night
* Alcohol abuse
* Regular use of sedatives
* Regular use of aspirin or cholesterol lowering agents

Study Group 2: Normal Controls

Inclusion Criteria:

* 21 years or older
* No diagnosis of intermittent hypoxemia (IH) or obstructive sleep apnea (OSA)
* No diagnosis of hypertension, coronary artery disease, diabetes, stroke, or evidence of underlying vascular disease

Exclusion Criteria:

* Smoking
* Pregnancy
* Known cardiovascular disease, stroke, or diabetes
* Use of supplemental oxygen at night
* Alcohol abuse
* Regular use of sedatives
* Regular use of aspirin or cholesterol lowering agents

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Krieger, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College - Weill Cornell Pulmonary Associates, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krieger AC, Anand R, Hernandez-Rosa E, Maidman A, Milrad S, DeGrazia MQ, Choi AJ, Oromendia C, Marcus AJ, Drosopoulos JHF. Increased platelet activation in sleep apnea subjects with intermittent hypoxemia. Sleep Breath. 2020 Dec;24(4):1537-1547. doi: 10.1007/s11325-020-02021-4. Epub 2020 Feb 8. PMID 32036486

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sleep Apnea | Normal Control
Started | 49 | 21
Completed | 49 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Apnea | Normal Control | Total
Number analyzed (Participants) | 49 | 21 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 21 | 68
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 43 | 15 | 58

OUTCOME MEASURES:

1. Primary Outcome: ODI
Description: The oxygen desaturation index (ODI) is the number of times per hour of sleep that the blood's oxygen level drop by a certain degree from baseline.
Time Frame: Day 1 (all subjects)
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Sleep Apnea | Normal Control
Number analyzed (Participants) | 49 | 21
events/hour | 24.71 (30.15) | .97 (1.43)

ADVERSE EVENTS:
Groups:
- Normal Control: Subject found to have no evidence of Obstructive Sleep Apnea (OSA) after Nocturnal Polysomnography (NPSG). These subjects will only undergo a blood draw and will not have the Continuous Positive Airway Pressure (CPAP) treatment.
  Serious and Other [Not Including Serious] Adverse Events were not observed.
- Sleep Apnea: Subjects found to have Obstructive Sleep Apnea (OSA) with Intermittent Hypoxemia (IH). This arm will undergo a pre-treatment blood draw, one month of Continuous Positive Airway Pressure (CPAP) to treat OSA, and a post-treatment blood draw.
  Continuous Positive Airway Pressure (CPAP): Continuous positive airway pressure (CPAP) is a method of respiratory ventilation which is accepted as the gold standard to treat Obstructive Sleep Apnea (OSA). Subjects found to have OSA after the Nocturnal Polysomnography (NPSG) will be trained in the use of CPAP and will be instructed to use CPAP every night for 30 nights. These subjects will then return for a post-treatment blood draw.
  Serious and Other [Not Including Serious] Adverse Events were not observed.
Arm/Group | Normal Control | Sleep Apnea
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/49
Other Adverse Events (participants affected / at risk) | 0/21 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes